CLINICAL TRIAL: NCT06473090
Title: Comparison of Using a Video vs. Text to Improve Learning of Secure Communication During a Crisis in Anesthesia: A Multicenter Randomized Controlled Study in Simulation
Brief Title: Comparison of Using a Video vs. a Text to Improve Secure Communication During a Crisis in Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Paris-Sud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LabForSims-007
Record Dates: First submitted 2024-06-12; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Simulation; Education; Communication
Keywords: Communication; education; simulation; anesthesia; video
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Parallel assignment, blinded, randomized study
Who Masked: Outcomes Assessor
Masking Description: The evaluation will be based on video recordings of the 2 scenarios assessed by 2 independent, blinded experts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Participants will watch a 15-minute educational video at the beginning of the session before their involvement in the 2 high-fidelity simulation scenarios.
  The educational video used was developed by experts (in Human Factors and Obstetric Anesthesia) and validated by SFAR and CARO. It depicts poor use of NTS (including CLC) during a maternal cardiac arrest anesthesia scenario and then proper use of NTS during the same scenario.
  Interventions: Other: Video group
- Text group (Active Comparator): Participants will read a text-type educational support for 15 minutes at the beginning of the session before their involvement in 2 high-fidelity crisis simulation scenarios.
  The text-type educational support, written in French by the same team of experts, covers all the NTS mentioned in the video and has already been used in a previous study
  Interventions: Other: Text group

INTERVENTIONS:
Other: Video group — Participants will watch a 15-minute educational video at the beginning of the session before their involvement in the 2 high-fidelity simulation scenarios.
  The educational video used was developed by experts (in Human Factors and Obstetric Anesthesia) and validated by SFAR and CARO. It depicts poor use of NTS (including CLC) during a maternal cardiac arrest anesthesia scenario and then proper use of NTS during the same scenario.
  Arms: Video group
Other: Text group — Participants will read a text-type educational support for 15 minutes at the beginning of the session before their involvement in 2 high-fidelity crisis simulation scenarios.
  The text-type educational support, written in French by the same team of experts, covers all the NTS mentioned in the video and has already been used in a previous study
  Arms: Text group

SUMMARY:
Poor team communication in the OR is associated with increased postoperative morbidity and mortality. Thus, experts recommend that the healthcare team in a crisis situation use secure and standardized communication to improve the quality and safety of care. Secure and standardized communication involves clear, concise, and unambiguous language. Methods of secure communication include closed-loop communication (CLC), precise and complete communication (direct, full dosage), and the use of the SBAR tool. To improve healthcare professionals' communication, it is essential to use effective educational tools. Traditionally, lectures or reading articles were the standard methods. The use of video as a tool for knowledge and skills transfer seems promising. The objective is to compare the learning of secure communication in crisis situations in anesthesia after using two different educational supports: a text versus an educational video.

A prospective, multicenter, controlled, and randomized study will be conducted during high-fidelity simulation sessions in anesthesia, comparing a group using a text-type educational support versus a group using an educational video. It will take place in simulation centers. Voluntary participants will be anesthesia and critical care residents and/or nurse anesthetists who have used one of the educational supports and then actively participated in the simulation scenarios. After their consent, participants will be randomized into two groups:

* Text group: Participants will read a text-type educational support for 15 minutes at the beginning of the session before their involvement in 2 high-fidelity crisis simulation scenarios.
* Video group: Participants will watch a 15-minute educational video at the beginning of the session before their involvement in the 2 high-fidelity simulation scenarios.

The primary endpoint will be to compare the total number of correct secure communication events during the crisis between the 2 groups, which includes: a) Number of correctly performed SBAR b) Number of correctly or partially performed closed-loop communications (CLC) c) Number of directive verbal orders d) Number of correct medication dosages. This evaluation will be based on video recordings of the 2 scenarios assessed by 2 independent, blinded experts (external evaluation of a team's secure communication skills (Kirkpatrick level 2). This composite score is based on various secure communication methods described in the literature and recommended by experts. The number of verbal orders per scenario will also be recorded.

The secondary endpoint will be to evaluate each item independently, the proportion of CLC per verbal order, satisfaction with the educational tool (Kirkpatrick level 1), and the perception of learning in terms of secure communication (1 to 10 Likert scale, Kirkpatrick level 2). Participants' characteristics will also be collected.

DETAILED DESCRIPTION:
Introduction Effective resolution of a crisis situation in anesthesia and critical care requires both technical and non-technical skills (1). Non-technical skills (NTS) include leadership, task distribution, teamwork, and communication. Moreover, communication issues are common in the operating room (2). Poor team communication in the OR is associated with increased postoperative morbidity and mortality (3). Thus, experts recommend that the healthcare team in a crisis situation use secure and standardized communication to improve the quality and safety of care (to reduce morbidity and mortality and limit the incidence of adverse events) (1). Secure and standardized communication involves clear, concise, and unambiguous language. Methods of secure communication include closed-loop communication (CLC), precise and complete communication (direct, full dosage), and the use of the SBAR tool (1).

To improve healthcare professionals' communication, it is essential to use effective educational tools. Traditionally, lectures or reading articles were the standard methods. More recently, simulation has shown its value in acquiring these skills (1)(4). However, given the large number of professionals and the limited number of trainers, other educational tools must be developed to allow training for as many professionals as possible.

The use of video as a tool for knowledge and skills transfer seems promising. Nowadays, many teenagers and adults regularly watch videos on digital platforms. Animated images offer many advantages over text. Research in psychology shows that 93% of human communication is non-verbal (5). Additionally, the human brain deciphers different elements of an image simultaneously, whereas spoken or written language is decoded linearly and sequentially, which takes more time (5). Consequently, the use of images for knowledge transfer would be particularly relevant as learning is more effective when visual, oral, or written information is provided simultaneously rather than sequentially (5). In the healthcare field, using images related to written or spoken text has proven particularly effective for knowledge transmission (6). Illustrated text allows participants to develop more complex cognitive structures than those who do not benefit from images (7).

Objective: The objective of this study is to compare the learning of secure communication in crisis situations in anesthesia after using two different educational supports: a text versus an educational video.

Materials and Methods A prospective, multicenter, controlled, and randomized study will be conducted during high-fidelity simulation sessions in anesthesia, comparing a group using a text-type educational support versus a group using an educational video. It will take place in simulation centers. Voluntary participants will be anesthesia residents and/or nurse anesthetists who have used one of the educational supports and then actively participated in the simulation scenarios.

After their consent, participants will be randomized into two groups:

* Text group: Participants will read a text-type educational support for 15 minutes at the beginning of the session before their involvement in 2 high-fidelity crisis simulation scenarios.
* Video group: Participants will watch a 15-minute educational video at the beginning of the session before their involvement in the 2 high-fidelity simulation scenarios.

The educational video used was developed by experts (in Human Factors and Obstetric Anesthesia) and validated by SFAR and CARO. It depicts poor use of NTS (including CLC) during a maternal cardiac arrest anesthesia scenario and then proper use of NTS during the same scenario. The text-type educational support, written in French by the same team of experts, covers all the NTS mentioned in the video and has already been used in a previous study (1)(5).

The 2 high-fidelity simulation scenarios will be crisis scenarios in anesthesia promoting verbal orders and communication (including cardiac arrest, malignant hyperthermia...). They will serve as the evaluation basis. Each scenario will involve 2 to 3 learner participants (residents and/or nurse anesthetists). The first scenario will be followed by a debriefing focusing on technical skills, and the second scenario will be followed by a debriefing focusing on both technical and non-technical skills.

The primary endpoint will be to compare the total number of correct secure communication events during the crisis between the 2 groups, which includes: a) Number of correctly performed SBAR (1 correct event = 1 point) b) Number of correctly or partially performed closed-loop communications (CLC) (1 correct event = 1 point, partial = ½ point) c) Number of directive verbal orders (using a name or the pronoun "you") (1 correct event = 1 point) d) Number of correct medication dosages (medication with route of administration and dosage) (1 correct event = 1 point) This evaluation will be based on video recordings of the 2 scenarios assessed by 2 independent, blinded experts. This composite score is based on various secure communication methods described in the literature and recommended by experts (1). It corresponds to an external evaluation of a team's secure communication skills (Kirkpatrick level 2). The number of verbal orders per scenario will also be counted by the 2 experts. A correct closed-loop communication is defined as completing the following 3 steps: 1° the sender formulates the order / 2° the receiver acknowledges receipt of the message / 3° the sender closes the loop by verifying the message is correctly received. The verbal order is only the first step when the sender formulates the order aloud.

The secondary endpoint will be to evaluate each item independently, the proportion of CLC per verbal order, satisfaction with the educational tool (Kirkpatrick level 1), and the perception of learning in terms of secure communication (rated between 1 to 10 on a Likert scale, Kirkpatrick level 2). Participants' characteristics will also be collected via an online questionnaire right after the session.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia residents and/or nurse anesthetists who have used one of the educational supports and then actively participated in the simulation scenarios.

Exclusion Criteria:

* technical problem video
* declines active participation in the session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-26 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
communication events | 30 minutes by video after the end of the session by an external evaluator
  The primary endpoint will be to compare the total number of correct secure communication events during the crisis between the 2 groups, which includes: a) Number of correctly performed SBAR (1 correct event = 1 point) b) Number of correctly or partially performed closed-loop communications (CLC) (1 correct event = 1 point, partial = ½ point) c) Number of directive verbal orders (using a name or the pronoun "you") (1 correct event = 1 point) d) Number of correct medication dosages (medication with route of administration and dosage) (1 correct event = 1 point). This evaluation will be based on video recordings of the 2 scenarios assessed by 2 independent, blinded experts. This composite score is based on various secure communication methods described in the literature and recommended by experts (1). It corresponds to an external evaluation of a team's secure communication skills (Kirkpatrick level 2).

SECONDARY OUTCOMES:
Satisfaction | 1 minute and the end of the session by all residents
  to evaluate satisfaction with the educational tool ((rated between 1 to 10 on a Likert scale, Kirkpatrick level 1)
perception of learning | 1 minute and the end of the session by all residents
  the perception of learning in terms of secure communication (rated between 1 to 10 on a Likert scale, Kirkpatrick level 2).
Closed-loop-communication | 30 minutes by video after the end of the session by an external evaluator
  to evaluate the proportion of Closed loop communication per verbal order.
SBAR (situation, background, assessment, recommandation) tool | 30 minutes by video after the end of the session by an external evaluator
  to evaluate Number of correctly performed SBAR tool (1 correct event = 1 point)
closed-loop communication | 30 minutes by video after the end of the session by an external evaluator
  to evaluate Number of correctly or partially performed closed-loop communications ( correct event = 1 point, partial = ½ point)
verbal orders | 30 minutes by video after the end of the session by an external evaluator
  to evaluate Number of directive verbal orders (using a name or the pronoun "you") (1 correct event = 1 point)
medication dosages | 30 minutes by video after the end of the session by an external evaluator
  d) Number of correct medication dosages (medication with route of administration and dosage) (1 correct event = 1 point).

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Blanié, MD PhD, Principal Investigator — Université Paris-Saclay

IPD SHARING:
Plan to Share IPD: No